CLINICAL TRIAL: NCT04103242
Title: Difference in Relative Abundance of Lactobacillus in Endometrium With and Without Histologically Proven Chronic Endometritis
Brief Title: Abundance of Lactobacillus in Endometrium Affected by Chronic Endometritis
Acronym: endoMB
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-01064 endoMB
Record Dates: First submitted 2018-10-31; First posted 2019-09-25 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Non Specific Chronic Endometritis; Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — endometrial samples swabs from Cervix uteri, vagina and uterine cavity
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 16s rRNA gene sequencing — High-throughput sequencing of the microbial 16s rRNA subunit to define the abundance of microbial phyla and genera

SUMMARY:
Infertile women undergoing hysteroscopy for diagnostic or therapeutic indication are asked to donate a sample of endometrium.

Endometrial samples of study participants are examined for signs of chronic endometritis by immunohistochemical analysis.

High-throughput sequencing of the microbial 16s ribosomal ribonucleic acid (rRNA) subunit is performed to identify and quantify the microbes present in the sample.

Obstetric and reproductive outcome is recorded 12 months after hysteroscopy (telephone interview).

ELIGIBILITY:
Inclusion Criteria:

* Infertile (≥ 12 months of unprotected regular intercourse) premenopausal women or women with ≥ 2 consecutive miscarriages undergoing hysteroscopy. - Infertile women undergoing office hysteroscopy for other reasons, such as suspected intrauterine adhesions after curettage, irregular endometrium, uterine polyps, repeated implantation failure in assisted reproduction, etc.
* Signed informed consent
* BMI ≥ 18 kg/m2 and ≤ 40 kg/m2
* Age: ≥ 18 years and ≤ 45 years
* follicle stimulating hormone (FSH) ≤ 20 (day 2-5 and estradiol ≤ 300 pmol/l)

Exclusion Criteria:

* Treatment with antibiotics in the past 3 months
* Treatment with immune-suppressing or immune-modulating drugs in the past 3 months
* Treatment with estrogens, progestins, contraceptives and/or antiestrogenic drugs in the cycle during which hysteroscopy is performed
* Current infection of the cervix with Chlamydia trachomatis and/or gonorrhea
* Pelvic surgery in the past 3 months
* Suspicion of malignancy
* Pregnancy
* Breast feeding
* Perimenopause (irregular menses and FSH ≥ 20 U/l on day 3-5 of the cycle)
* Outdated endometrial sample from the luteal phase (this criterion will be evaluated during visit 4 post surgery)
* Elevated progesterone concentration ≥ 20 nmol/l measured in the blood sample taken at the time of HSC.
* Insufficient amount of tissue for immunohistochemical analysis and/or microbial 16s rRNA gene sequencing

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients presenting at the Clinic for Reproductive Medicine of the University Hospital Basel because of infertility with an indication for HSC represent the project population.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Quantity of Lactobacillus | 1 year
  Quantity of Lactobacillus determined by 16S ribosomal RNA gene sequencing
alpha diversity of microbes | 1 year
  Quantification of microbes and their diversity within the individual endometrium sample
Shannon index (Beta diversity) | 1 Year
  Comparison of microbial diversity among the subjects

SECONDARY OUTCOMES:
Pregnancy Rate | 2 years
  Number of pregnancies within 12 months after hysteroscopy
Live Birth Rate | 3 years
  Number of pregnancies within 12 months after hysteroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Moffat, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No